CLINICAL TRIAL: NCT02964377
Title: A Single Center Dose Ranging Pilot Study of (+)-Epicatechin in Non-ambulatory Adolescents With Duchenne Muscular Dystrophy and Pre-symptomatic Cardiac Dysfunction
Brief Title: Plus Epicatechin Duchenne Muscular Dystrophy in Non-ambulatory Adolescents
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Craig McDonald, MD (Other)
Collaborators: Cardero Therapeutics, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Craig McDonald, MD, Professor and Chair of Department of Physical Rehabilitation, University of California, Davis
Organization: University of California, Davis (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 951753
Record Dates: First submitted 2016-11-07; First posted 2016-11-16 (Estimated); Results first posted 2021-12-21 (Actual); Last update posted 2021-12-21 (Actual); Status verified 2021-11

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Pediatric; muscle disease; Duchenne muscular dystrophy; cardiomyopathy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Muscular Diseases; Cardiomyopathies | interventions — Catechin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cohort 1 (Experimental): 8-weeks open-label (+)- Epicatechin at 25mg/day twice per day,
  Interventions: Drug: (+)- Epicatechin
- Cohort 2 (Experimental): 8-weeks open-label (+)- Epicatechin at 25mg/day three times per day
  Interventions: Drug: (+)- Epicatechin
- Cohort 3 (Experimental): 8-weeks open-label (+)- Epicatechin at 75mg/day at two times per day
  Interventions: Drug: (+)- Epicatechin

INTERVENTIONS:
Drug: (+)- Epicatechin

SUMMARY:
This single center open-label pilot study will enroll 15 non-ambulatory children with Duchenne muscular dystrophy at least 8 years of age and who demonstrate pre-clinical cardiomyopathy (defined as a cardiac ejection fraction >55% with abnormal LV strain by cardiac MRI). They will receive (+)-epicatechin at one of three doses during an 8-week dose-ranging study with assessments at baseline, 2 Weeks, 4weeks, and 8 weeks. The study will determine optimal dosing for future cardiac efficacy studies based on serum / plasma biomarker response using follistatin: myostatin ratio, nitrite/nitrate ratio, cardiac troponins and cardiac BNP. Secondary endpoints will include additional biomarker assessments by SOMAscanTM, cardiac functional evaluations by cardiac MRI (LV strain), and echocardiogram (LV strain by speckle tracking) and measures of strength, range of motion and mobility, and clinical safety assessments. Results of secondary endpoint analysis will be used to refine design of subsequent clinical trials powered to detect changes in clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Age 8 years to 17 years
* Non-Ambulatory (unable to complete 10m run/walk under 10s)
* Weight </=100Kg
* Diagnosis of DMD confirmed by at least one the following:

  * Dystrophin immunofluorescence and/or immunoblot showing complete dystrophin deficiency, and clinical picture consistent with typical DMD, or
  * Gene deletions test positive (missing one or more exons) of the dystrophin gene, where reading frame can be predicted as 'out-of-frame', and clinical picture consistent with typical DMD, or
  * Complete dystrophin gene sequencing showing an alteration (point mutation, duplication, or other mutation resulting in a stop codon mutation) that can be definitely associated with DMD, with a typical clinical picture of DMD, or
  * Positive family history of DMD confirmed by one of the criteria listed above in a sibling or maternal uncle, and clinical picture typical of DMD.
* Cardiac ejection fraction >55% on echocardiogram
* Use of nutritional, herbal and antioxidant supplements taken with the intent of maintaining or improving skeletal muscle strength or functional mobility has been discontinued at least 4 weeks prior to screening (daily multivitamin use is acceptable).
* Glucocorticoid therapy, if used, must have a stable weight-based dose for at least 3 months prior to enrollment
* Cardiac therapy, if used, includes prophylactic ACE inhibitors, aldosterone receptor antagonists (e.g.

spironolactone, eplerenone, etc.), and/or beta-blocker therapy, and must be stable for 3 months prior to enrollment.

* Hematology profile within normal range.
* Baseline laboratory safety chemistry profile within typical range for DMD (elevated ALT / AST acceptable in the absence of elevated GGT, elevated CK acceptable).

Exclusion Criteria:

* Inability to complete cardiac or strength, range of motion and mobility assessments per protocol
* Current enrollment in another treatment clinical trial.
* History of significant concomitant illness or significant impairment of renal or hepatic function.
* Use of regular daily aspirin or other medication with antiplatelet effects within 3 weeks of first dose of study medication.
* Cardiac symptoms that, in the opinion of the investigator, may be suggestive of imminent moderate to severe cardiac events, irrespective of LVEF.

Ages: 8 Years to 17 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UC Davis Medical Center, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: (+)- Epicatechin at 25mg/day twice per day
- Cohort 2: (+)- Epicatechin at 25mg/day three times per day
- Cohort 3: (+)- Epicatechin at 75mg/day at two times per day.
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Started | 5 | 5 | 5
Completed | 5 | 5 | 5
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Total
Number analyzed (Participants) | 5 | 5 | 5 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.2 (3.1) | 11.9 (3.0) | 13.2 (2.9) | 12.8 (2.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 5 | 5 | 5 | 15
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics Outcome: Absolute Values of (+)-Epicatechin Serum Concentration, Pre-dose (Trough) and 2 Hours Post-dose (Peak)
Description: Pharmacokinetic evaluation for dose-response evaluation.
Time Frame: Pre-dose and 2 hours post-dose at baseline
Population: One Cohort 3 participant post-dose sample was missed.
Measure: Mean (Standard Deviation); unit: nM
Groups:
- Cohort 1: 8-weeks open-label (+)- Epicatechin at 25mg/day twice per day
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 5 | 5 | 4
nM
  Trough | 15.1 (10.4) | 33.9 (7.9) | 20.6 (43.6)
  Peak | 481.2 (477.6) | 551.2 (284.9) | 3899.3 (1217.6)
Statistical Analysis 1: Comparison: Cohort 1; Test type: Equivalence — Difference in trough vs. peak values was evaluated using a paired t-test analysis; p = 0.0482, t-test, 2 sided
Statistical Analysis 2: Comparison: Cohort 2; Test type: Equivalence — Difference in trough vs. peak values was evaluated using a paired t-test analysis; p = 0.0075, t-test, 2 sided
Statistical Analysis 3: Comparison: Cohort 3; Test type: Equivalence — Difference in trough vs. peak values was evaluated using a paired t-test analysis; p = 0.0083, t-test, 2 sided

2. Primary Outcome: Pharmacokinetics Outcome: Absolute Values of (+)-Epicatechin Serum Concentration, Pre-dose (Trough) and 2 Hours Post-dose (Peak)
Description: Pharmacokinetic evaluation for dose-response evaluation.
Time Frame: Week 4
Measure: Mean (Standard Deviation); unit: nM
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 5 | 5 | 5
nM
  Trough | 84.2 (47.6) | 163.8 (84.5) | 179.1 (398.1)
  Peak | 742.8 (442.7) | 601 (357) | 5590.8 (1729.9)
Statistical Analysis 1: Comparison: Cohort 1; Test type: Equivalence — Difference in trough vs. peak values was evaluated using a paired t-test analysis; p = 0.0127, t-test, 2 sided
Statistical Analysis 2: Comparison: Cohort 2; Test type: Equivalence — Difference in trough vs. peak values was evaluated using a paired t-test analysis; p = 0.0202, t-test, 2 sided
Statistical Analysis 3: Comparison: Cohort 3; Test type: Equivalence — Difference in trough vs. peak values was evaluated using a paired t-test analysis; p = 0.0007, t-test, 2 sided

3. Primary Outcome: Laboratory Outcome: Absolute Plasma Follistatin:Myostatin Ratio at Baseline, Week 4 and Week 8
Description: Evaluation of follistatin:myostatin ratio from plasma samples.
Time Frame: Baseline, Week 4 and Week 8
Measure: Mean (Standard Deviation); unit: Ratio of follistatin to myostatin (AU)
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 5 | 5 | 5
Ratio of follistatin to myostatin (AU)
  Baseline | 1.82 (0.71) | 1.76 (0.74) | 3.31 (0.91)
  Week 4 | 3.61 (0.78) | 3.41 (1.24) | 5.26 (0.87)
  Week 8 | 4.02 (1.55) | 3.94 (1.23) | 5.7 (0.65)
Statistical Analysis 1: Comparison: Cohort 1; Baseline vs. Week 4 (Cohort 1); Test type: Other — Mixed Model Repeated Measures (MMRM) regression; p < 0.0001, Regression, Linear
Statistical Analysis 2: Comparison: Cohort 2; Baseline vs. Week 4 (Cohort 2); Test type: Other — Mixed Model Repeated Measures (MMRM) regression; p < 0.0001, Regression, Linear
Statistical Analysis 3: Comparison: Cohort 3; Baseline vs. Week 4 (Cohort 3); Test type: Other — Mixed Model Repeated Measures (MMRM) regression; p < 0.0001, Regression, Linear
Statistical Analysis 4: Comparison: Cohort 1; Baseline vs. Week 8 (Cohort 1); Test type: Other — Mixed Model Repeated Measures (MMRM) regression; p < 0.0001, Regression, Linear
Statistical Analysis 5: Comparison: Cohort 2; Baseline vs. Week 8 (Cohort 2); Test type: Other — Mixed Model Repeated Measures (MMRM) regression; p < 0.0001, Regression, Linear
Statistical Analysis 6: Comparison: Cohort 3; Baseline vs. Week 8 (Cohort 3); Test type: Other — Mixed Model Repeated Measures (MMRM) regression; p < 0.0001, Regression, Linear

4. Primary Outcome: Clinical Outcome: Mean Percent of Baseline Cardiac Ejection Fraction by MRI
Description: Evaluation of change in cardiac volume and performance, as measured by the mean percent of baseline ejection fraction using Cardiac MRI, measured at 8 weeks.
Time Frame: Week 8
Population: Missing data due to poor image quality.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 4 | 5 | 2
percentage | 98.19 (14.92) | 96.23 (9.66) | 92.27 (14.98)

5. Primary Outcome: Safety: Number of Participants Who Experienced Treatment-Related Laboratory Abnormalities
Description: Treatment-related laboratory abnormalities, defined as values outside of the typical range for Duchenne Muscular Dystrophy. Safety laboratory tests included blood chemistry panel, complete blood count w/ differential panel, & urinalysis assessments for clinical safety monitoring.
Time Frame: Study duration (8 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 5 | 5 | 5
Participants | 1 | 0 | 2

6. Primary Outcome: Laboratory Outcome: Absolute Values of Nitric Oxide (AU) Measured by ELISA
Description: Proteomics evaluation of plasma biomarkers to confirm intervention-responsive pathophysiological pathways, using enzyme-linked immunosorbent assay (ELISA).
Time Frame: Baseline, Week 4, Week 8
Measure: Mean (Standard Deviation); unit: AU
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 5 | 5 | 5
AU
  Baseline | 0.65 (0.17) | 0.63 (0.14) | 0.57 (0.21)
  Week 4 | 0.82 (0.31) | 1.06 (0.16) | 0.93 (0.36)
  Week 8 | 0.99 (0.28) | 1.14 (0.15) | 0.92 (0.3)
Statistical Analysis 1: Comparison: Cohort 1; Baseline vs. Week 4; Test type: Other — Mixed Model Repeated Measures (MMRM) regression; p = 0.002, Regression, Linear
Statistical Analysis 2: Comparison: Cohort 2; Baseline vs. Week 4; Test type: Other — Mixed Model Repeated Measures (MMRM) regression; p < 0.001, Regression, Linear
Statistical Analysis 3: Comparison: Cohort 3; Baseline vs. Week 4; Test type: Other — Mixed Model Repeated Measures (MMRM) regression; p < 0.0001, Regression, Linear
Statistical Analysis 4: Comparison: Cohort 1; Baseline vs. Week 8; Test type: Other — Mixed Model Repeated Measures (MMRM) regression; p < 0.0001, Regression, Linear
Statistical Analysis 5: Comparison: Cohort 2; Baseline vs. Week 8; Test type: Other — Mixed Model Repeated Measures (MMRM) regression; p < 0.0001, Regression, Linear
Statistical Analysis 6: Comparison: Cohort 3; Baseline vs. Week 8; Test type: Other — Mixed Model Repeated Measures (MMRM) regression; p < 0.0001, Regression, Linear

7. Primary Outcome: Laboratory Outcome: Absolute Values of Carbonylation (AU) Measured by ELISA
Description: as for outcome 6
Time Frame: Baseline, Week 4, Week 8
Measure: Mean (Standard Deviation); unit: AU
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 5 | 5 | 5
AU
  Baseline | 12.85 (2.38) | 15.7 (1.74) | 12.45 (3.91)
  Week 4 | 9.95 (1.72) | 12.2 (2.08) | 7.18 (2.74)
  Week 8 | 9.07 (1.41) | 10.47 (1.91) | 6.64 (1.05)
Statistical Analysis 1: Comparison: Cohort 1; Baseline vs. Week 4; Test type: Other — Mixed Model Repeated Measures (MMRM) regression; p < 0.0001, Regression, Linear
Statistical Analysis 2: Comparison: Cohort 2; Baseline vs. Week 4; Test type: Other — Mixed Model Repeated Measures (MMRM) regression; p < 0.0001, Regression, Linear
Statistical Analysis 3: Comparison: Cohort 3; Baseline vs. Week 4; Test type: Other — Mixed Model Repeated Measures (MMRM) regression; p < 0.0001, Regression, Linear
Statistical Analysis 4: Comparison: Cohort 1; Baseline vs. Week 8; Test type: Other — Mixed Model Repeated Measures (MMRM) regression; p < 0.0001, Regression, Linear
Statistical Analysis 5: Comparison: Cohort 2; Baseline vs. Week 8; Test type: Other — Mixed Model Repeated Measures (MMRM) regression; p < 0.0001, Regression, Linear
Statistical Analysis 6: Comparison: Cohort 3; Baseline vs. Week 8; Test type: Other — Mixed Model Repeated Measures (MMRM) regression; p < 0.0001, Regression, Linear

8. Primary Outcome: Laboratory Outcome: Absolute Values of Follistatin (AU) Measured by ELISA
Description: as for outcome 6
Time Frame: Baseline, Week 4, Week 8
Measure: Mean (Standard Deviation); unit: AU
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 5 | 5 | 5
AU
  Baseline | 527.24 (282.06) | 555.71 (382.28) | 1011.25 (247.39)
  Week 4 | 891.43 (278.51) | 795.71 (352.83) | 1356.25 (117.13)
  Week 8 | 951.43 (312.39) | 914.29 (350.17) | 1351.25 (148.95)
Statistical Analysis 1: Comparison: Cohort 1; Baseline vs. Week 4; Test type: Other — Mixed Model Repeated Measures (MMRM) regression; p < 0.0001, Regression, Linear
Statistical Analysis 2: Comparison: Cohort 2; Baseline vs. Week 4; Test type: Other — Mixed Model Repeated Measures (MMRM) regression; p < 0.0001, Regression, Linear
Statistical Analysis 3: Comparison: Cohort 3; Baseline vs. Week 4; Test type: Other — Mixed Model Repeated Measures (MMRM) regression; p < 0.0001, Regression, Linear
Statistical Analysis 4: Comparison: Cohort 1; Baseline vs. Week 8; Test type: Other — Mixed Model Repeated Measures (MMRM) regression; p < 0.0001, Regression, Linear
Statistical Analysis 5: Comparison: Cohort 2; Baseline vs. Week 8; Test type: Other — Mixed Model Repeated Measures (MMRM) regression; p < 0.0001, Regression, Linear
Statistical Analysis 6: Comparison: Cohort 3; Baseline vs. Week 8; Test type: Other — Mixed Model Repeated Measures (MMRM) regression; p < 0.0001, Regression, Linear

9. Primary Outcome: Laboratory Outcome: Absolute Values of Myostatin (AU) Measured by ELISA
Description: as for outcome 6
Time Frame: Baseline, Week 4, Week 8
Measure: Mean (Standard Deviation); unit: AU
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 5 | 5 | 5
AU
  Baseline | 282.33 (69.7) | 302.33 (91.15) | 316.6 (88.7)
  Week 4 | 247.67 (66.94) | 239 (90.2) | 263.67 (56.16)
  Week 8 | 247.07 (69.7) | 233.67 (78.47) | 241.67 (51.67)
Statistical Analysis 1: Comparison: Cohort 1; Baseline vs. Week 4; Test type: Other — Mixed Model Repeated Measures (MMRM) regression; p = 0.012, Regression, Linear
Statistical Analysis 2: Comparison: Cohort 2; Baseline vs. Week 4; Test type: Other — Mixed Model Repeated Measures (MMRM) regression; p < 0.0001, Regression, Linear
Statistical Analysis 3: Comparison: Cohort 3; Baseline vs. Week 4; Test type: Other — Mixed Model Repeated Measures (MMRM) regression; p < 0.0001, Regression, Linear
Statistical Analysis 4: Comparison: Cohort 1; Baseline vs. Week 8; Test type: Other — Mixed Model Repeated Measures (MMRM) regression; p = 0.01, Regression, Linear
Statistical Analysis 5: Comparison: Cohort 2; Baseline vs. Week 8; Test type: Other — Mixed Model Repeated Measures (MMRM) regression; p < 0.0001, Regression, Linear
Statistical Analysis 6: Comparison: Cohort 3; Baseline vs. Week 8; Test type: Other — Mixed Model Repeated Measures (MMRM) regression; p < 0.0001, Regression, Linear

10. Secondary Outcome: Clinical Outcome: Percent of Normalized Upper Extremity Reachable Surface Area at Week 4 and Week 8
Description: Quantitative upper extremity reachable workspace will be assessed using the XBox Kinect system. The KINECT Upper Extremity Reachable Workspace test measures surface area of a reachable workspace "bubble", normalized to the size of the individual, noted as the RSA or Reachable Surface Area. The Total RSA measure is the sum of four quadrants dividing superior and inferior medial and lateral spaces. A total score of 1 indicates a typical reachable workspace, while lower scores indicate restrictions in one or more of the four quadrants.
Time Frame: Baseline, Week 4, Week 8
Population: Missing data due to equipment malfunction
Measure: Mean (Standard Deviation); unit: % normalized reachable surface area
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 4 | 5 | 4
% normalized reachable surface area
  Baseline | 44 (33.9) | 89.9 (24.6) | 33 (23.2)
  Week 4: number analyzed (Participants) | 3 | 5 | 4
  Week 4 | 63.7 (44.4) | 84.4 (32.9) | 35.8 (21.4)
  Week 8 | 47.9 (51.2) | 92.7 (35.4) | 41.5 (26.7)

11. Secondary Outcome: Clinical Outcome: Total Score Using Performance of the Upper Limb Assessment
Description: The standardized Performance of Upper Limb (PUL) measure will be assessed at baseline and after 4 & 8 weeks.
  The Performance of the Upper Limb module is an observer-administered performance battery of upper extremity mobility tasks for the shoulder (upper, 6 items, 12 points), elbow (middle, 9 items, 17 points) and wrist/hand (distal, 7 items, 13 points). Higher scores indicate higher level of function. Total score ranges from 0-42 points and is the sum of the scores for the three subscales (10 upper, 10 mid, and 14 distal).
Time Frame: Baseline, Week 4, Week 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 5 | 5 | 5
score on a scale
  Baseline | 19.8 (5.4) | 30.8 (6.8) | 27 (10.6)
  Week 4 | 21.4 (6.8) | 32 (5.8) | 26.8 (9.9)
  Week 8 | 22 (5.8) | 31.8 (5.4) | 25.6 (11.4)
Statistical Analysis 1: Comparison: Cohort 1; Baseline vs. Week 4; Test type: Other — Mixed Model Repeated Measures (MMRM) regression; p = 0.01, Regression, Linear
Statistical Analysis 2: Comparison: Cohort 2; Baseline vs. Week 4; Test type: Other — Mixed Model Repeated Measures (MMRM) regression; p = 0.019, Regression, Linear
Statistical Analysis 3: Comparison: Cohort 1; Baseline vs. Week 8; Test type: Other — Mixed Model Repeated Measures (MMRM) regression; p < 0.001, Regression, Linear
Statistical Analysis 4: Comparison: Cohort 2; Baseline vs. Week 8; Test type: Other — Mixed Model Repeated Measures (MMRM) regression; p = 0.05, Regression, Linear

12. Secondary Outcome: Clinical Outcome: Mean Maximal Attained Revolutions Per 6-minute Cycle Test
Description: The Assisted Six-Minute Cycle Test is an ergometer-based assessment of upper limb function. Test results indicate the maximum number of ergometer revolutions achieved in six-minutes, with higher numbers indicating a greater degree of functional capacity.
Time Frame: Baseline, Week 4, Week 8
Measure: Mean (Standard Deviation); unit: revolutions
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 5 | 5 | 5
revolutions
  Baseline | 177.4 (112.4) | 362.6 (82.8) | 330.8 (172.5)
  Week 4 | 194.4 (80.4) | 415 (77.2) | 348.2 (222.3)
  Week 8 | 199 (96.6) | 387 (54) | 356.8 (275.4)
Statistical Analysis 1: Comparison: Cohort 1; Baseline vs. Week 8; Test type: Other — Mixed Model Repeated Measures (MMRM) regression; p = 0.054, Regression, Linear — p-value for difference at Week 4
Statistical Analysis 2: Comparison: Cohort 2; Baseline vs. Week 4; Test type: Other — Mixed Model Repeated Measures (MMRM) regression; p = 0.009, Regression, Linear

13. Secondary Outcome: Person-Reported Outcome: Upper Extremity Standardized Mean Score Using Pediatric Outcomes Data Collection Instrument (PODCI) Quality of Life Instrument
Description: The PODCI instrument was developed by Daltroy and colleagues with support by the Pediatric Orthopaedic Society of North America (POSNA). The PODCI is a 108-item questionnaire that evaluates global functioning in the pediatric orthopedic population utilizing four components: upper extremity functioning, transfers and basic mobility, sports and physical functioning and a comfort/pain score. Global functioning is assessed by the average of the four previous scores. All scales are scored from zero to 100, with 100 representing the highest level of functioning and least pain. The PODCI asks questions such as "During the last week, was it easy or hard for you to … lift heavy books".
Time Frame: Baseline to Week 4 and Week 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 5 | 5 | 5
score on a scale
  Baseline | 32 (12.9) | 62.6 (24.6) | 66 (22.3)
  Week 4 | 31.2 (16.4) | 74.6 (18.3) | 72.6 (21.3)
  Week 8 | 36.2 (12.3) | 71 (21.6) | 62.6 (32.1)
Statistical Analysis 1: Comparison: Cohort 1; Baseline vs. Week 8; Test type: Other — Mixed Model Repeated Measures (MMRM) regression; p = 0.025, Regression, Linear
Statistical Analysis 2: Comparison: Cohort 2; Baseline vs. Week 4; Test type: Other — Mixed Model Repeated Measures (MMRM) regression; p = 0.026, Regression, Linear

14. Secondary Outcome: Person-Reported Outcome: Mean Person-Reported Outcome Measure Upper Limb (PROM-UL) Functional Capacity Score
Description: The Performance of Upper Limb module (PUL) for DMD was designed according to a specific contextual framework of upper limb function in both ambulant and non-ambulant individuals with DMD. The UL-PROM closely linked to this motor performance based clinician-reported outcome measure, was developed to evaluate manual ability related to activities of daily living (ADL) that cannot be observed in a clinical setting. Items were selected in relation to the different domains of the PUL from proximal to distal performance in order to cover the full range of upper limb functions. The questionnaire consists of 33 items covering four domains (3 points each for Food/Nutrition 7 items, Self Care 8 items, Household/Environment 6 items, Leisure/Communication 12 items). Higher scores indicate greater function, with total score being a sum of the subscale scores (Ranging from 0 to 99).
Time Frame: Change from Baseline to Week 4 and Week 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 5 | 5 | 5
score on a scale
  Baseline | 73.6 (19.8) | 88.4 (7.9) | 79.2 (24.1)
  Week 4 | 64 (14.5) | 87.4 (7.6) | 82.8 (20.2)
  Week 8 | 62.6 (15) | 87.6 (6.3) | 78.8 (18.5)
Statistical Analysis 1: Comparison: Cohort 1; Baseline vs. Week 4; Test type: Other — Mixed Model Repeated Measures (MMRM) regression; p = 0.006, Regression, Linear
Statistical Analysis 2: Comparison: Cohort 1; Baseline vs. Week 8; Test type: Other — Mixed Model Repeated Measures (MMRM) regression; p = 0.002, Regression, Linear

15. Other Pre Specified Outcome: Clinical Outcome: Mean Strain Index (Ecc%) of Cardiac Mid-Ventricular Strain by MRI
Description: Cardiac MRI using tagged imaging detects changes in heart muscle contractility in people with DMD. It measures how the heart deforms throughout the cardiac cycle, and is used to calculate strain on the heart muscle. Peak strain is a measure of distortion in the heart muscle during contraction versus when it is at rest. Mid-ventricular peak circumferential strain is a sensitive marker of cardiac function and can detect effects of therapeutic interventions. Strain is expressed in the negative, so more negative measurements indicate a healthy state while less negative measurements (closer to zero) indicate an unhealthy state.
Time Frame: Baseline, Week 8
Population: 3 of the participants were unable to undergo the procedure and thus were not included in the analysis.
Measure: Mean (Standard Deviation); unit: Ecc%
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 5 | 4 | 3
Ecc%
  Baseline | -16.65 (4.31) | -17.38 (2.17) | -11.46 (1.34)
  Week 8 | -16.8 (1.39) | -17.67 (2.9) | -10.71 (6.0)

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 4/5 | 2/5 | 4/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=5) | Cohort 2 (N=5) | Cohort 3 (N=5)
Headache (General disorders) | 2 (3) | 0 (0) | 3 (5)
Stomach upset (General disorders) | 0 (0) | 0 (0) | 1 (1)
Troponin elevation (Cardiac disorders) | 0 (0) | 1 (2) | 3 (4)
Seasonal cold (General disorders) | 2 (2) | 1 (1) | 1 (1)
Sinus congestion (General disorders) | 1 (1) | 0 (0) | 0 (0)
Skin rash (diaper rash) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea/vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Strep throat (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Flu-like symptoms (General disorders) | 0 (0) | 0 (0) | 1 (1)
Cough, lower respiratory congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Body aches (General disorders) | 0 (0) | 0 (0) | 1 (1)
Vision, diagnosed as needing glasses (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Elevated triglycerides (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-11-14): https://cdn.clinicaltrials.gov/large-docs/77/NCT02964377/Prot_SAP_000.pdf
  • Informed Consent Form (2017-02-09): https://cdn.clinicaltrials.gov/large-docs/77/NCT02964377/ICF_001.pdf